CLINICAL TRIAL: NCT04182269
Title: Reliability and Validity of the Glittre Activities of Daily Living Test in Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gözde KAYA, Research Assistant, Hacettepe University
Other Study IDs: Hacettepe UN
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Glittre ADL test; Functional capacity assesment
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Multiple Sclerosis Patients
  Interventions: Other: Measurement of functional exercise capacity
- Control Group: Healthy Subjects
  Interventions: Other: Measurement of functional exercise capacity

INTERVENTIONS:
Other: Measurement of functional exercise capacity — The Glittre Activities of Daily Living (ADL) Test was used to evaluate functional exercise capacity.

SUMMARY:
Patients with Multiple Sclerosis (MS) have reduced functional capacity due to clinical symptoms of the disease, resulting in decreased participation in daily living activities and reduced quality of life. Evaluation of functional capacity and activities of daily living is very important in order to determine appropriate rehabilitation programs and increase the participation of patients in daily life activities. However, although there are many scales evaluating functional capacity and activities of daily living in people with disabilities, there is no specific assessment scale specific to MS patients. Therefore, this study was planned to investigate whether the Glittre Daily Living Activities (ADL) Test, which was developed to measure functional capacity in chronic obstructive pulmonary disease, is a valid and reliable measurement tool in MS patients. For this purpose, a total of 51 participants (25 MS patients and 26 healthy participants) evaluated with Glittre ADL Test.

The relationship between Glittre ADL Test and 6-minute walk test, Notthingham Extended Daily Living Activities Index, Multiple Sclerosis Quality of Life Scale, Fatigue Severity Scale, Balance Assessment Systems Test (MiniBEST Test), Extended Disability Status Scale and 5-repetition sit-to-stand test evaluated with Pearson or Spearman correlation coefficient. For the known group validity, the difference between the patient and control groups compared with the test of the difference between the two means. For reliability, test retest performed. Reliability evaluated with the intraclass correlation coefficient.

Hypothesis 1: Glittre ADL Test results in MS patients and healthy subjects are different.

Hypothesis 2: Glittre ADL Test is reliable in MS patients.

Hypothesis 3: Glittre ADL Test is valid for evaluating functional exercise capacity in MS patients.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic, inflammatory disease characterized by demyelination, myelin damage, axonal loss and gliosis in the Central Nervous System (CNS). MS symptoms vary according to the size of the lesion and its location in the CNS. Clinical symptoms are generally: spasticity, fatigue, muscle weakness, tremor, pain, sensory disturbances, bladder bowel problems, cognitive disorders, depression and sleep disorders. With the progression of the disease, the performance in daily living activities gradually decreases, affecting the quality of life negatively. Maintaining aerobic capacity in chronic diseases such as MS is very important for independence in daily living activities. Functional exercise capacity of MS patients decreases with the effect of symptoms and sedentary lifestyle. The decrease in aerobic capacity can manifest itself with a decrease in walking distance or speed, or a limitation in daily living activities. Decline in aerobic capacity is also associated with many factors such as increased risk of cardiovascular disease, decreased cognitive functions and health-related quality of life. Therefore, aerobic capacity measurement is one of the important physiological measurements in terms of evaluating the existing functional status of individuals and preparing rehabilitation programs appropriately for individuals.

Cardiopulmonary exercise tests (CPET) are accepted as the gold standard in the evaluation of aerobic capacity. These measurements have some limitations that limit their use, such as the high cost of equipment and the need for a well trained team. Today, submaximal tests, questionnaires or scales are widely used as an alternative to CPET in evaluating functional exercise capacity. Since most daily life activities are at the submaximal level, submaximal tests can better determine the functional levels of individuals in daily living activities.

In order to evaluate functional capacity in Chronic Obstructive Pulmonary Disease (COPD), activities similar to daily life activities were selected and the Glittre Daily Living Activities (ADL) Test was developed. It has been shown that the Glittre ADL Test is reliable and valid in evaluating functional exercise capacity in COPD, as well as reflecting the performance in daily living activities for this disease group. The activities in the Glittre ADL Test are those that require the use of both the lower and upper extremities. An important advantage of the test is that the test can reflect functional capacity as well as providing information about performance in daily life activities and that the use of all extremities can be observed during the test.

In this study, the reliability and validity of the Glittre ADL Test in MS patients was investigated. For the criterion validity of the Glittre ADL Test, the correlation with the 6-minute walk test (6MWT) was examined. Patient and control groups were compared for known group validity. Test-retest method was used to determine the reliability of Glittre ADL Test. Intra-observer reliability was evaluated by intraclass correlation coefficient (ICC). The relationship between Glittre ADL Test scores and lower extremity muscle strength, limitation of daily living activities, balance, quality of life, fatigue and disease severity was investigated. Correlations between the time to complete the Glittre ADL Test and the 5 Repetition Sit To Stand Test completion time, Nottingham Extended Activities of Daily Living Scale, Mini Balance Evulation Systems Test, Multiple Sclerosis Quality of Life 54 scale, Fatigue Severity Scale and Expanded Disability Status Scale scores were examined.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years
* Relapsing Remitting Multiple Sclerosis (RRMS) type MS disease.
* Extended Disability Status Scale (EDSS) score of maximum 4.5
* No attacks during the last 3 months
* The medication has not been changed in the last 6 months.
* Getting more than 24 points from the Standardized Mini Mental Test.

Exclusion Criteria

* Having had any musculoskeletal surgery.
* Using a walking aid or orthosis.
* Having a neurological disease other than MS.
* Having orthopedic or rheumatological problems that will affect function.
* Having a peripheral vestibular problem.
* Having a cardiovascular and pulmonary disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers of the patients who applied to Hacettepe University Neurology Department, diagnosed with MS by specialist physician and referred to Hacettepe University Faculty of Health Sciences Physiotherapy and Rehabilitation Department for physiotherapy and rehabilitation program were included in the study.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Glittre Activities of Dailiy Living Test | 10 minute
  Functional exercise capacity measurement

SECONDARY OUTCOMES:
6 minute walk test (6MWT) | 10 minute
  Functional exercise capacity measurement 6MWT was performed in accordance with American Thoracic Society guidelines. The start and end points of the test were determined. The test was carried out in a 30-meter corridor, avoiding distractions. 6-minute walking distance recorded in meters at the end of the test.
Nottingham Extended Daily Living Activities Index (NGGYAI) | 10 minute
  Nottingham Extended Daily Living Activities Index (NGGYAI) was used to evaluate the daily living activities. In addition to the Turkish validity and reliability of the index, it has been reported that it is reliable and valid in MS patients. The scale consists of 22 questions covering mobility, kitchen, home and entertainment activities. A higher score 0-66 scale indicates a better activities of daily living.
Extended Disability Status Scale (EDSS) | minimum 30 minute
  Expanded Disability Status Scale (EDSS) is the most commonly used scale to monitor disease stage and assess disability in multiple sclerosis patients.
  Eight functional systems (FS) are evaluated with EDSS (Visual functions, brain stem functions, pyramidal functions, cerebellar functions, sensory functions, bladder and bowel functions, cerebral functions and other). In addition, gait is also evaluated and a score between 0 (normal neurological status) and 10 (death due to MS) is determined by considering functional system scores and the level of independence of the patient in ambulation.
Fatigue Severity Scale | 10 minute
  Fatigue severity scale was used to evaluate the severity of fatigue. The scale consists of 9 items.
  Patients are asked to choose one of the options from 1 to 7 for each item in the scale.
  The Fatigue Severity Scale score is calculated by averaging the scores of the answers given to the nine items. A high score indicates an increase in the severity of fatigue.
Multiple Sclerosis Quality of Life İnstrument - 54 (MSQOL-54) | 15 minute
  Multiple sclerosis quality of life instrument (MSQOL-54), which was developed for MS patients and was validated and reliable in Turkish, was used to evaluate the quality of life of the patients.
  The scale consists of 14 subheading and 54 items. Each subheading is evaluated out of 100 points and 100 points represent the best status and 0 points represent the worst.
  The scores of the patients according to their answers to each question are calculated under 14 subheading.
  Then, with a separate calculation, according to the scores obtained from 14 subheading, 2 separate scores are obtained as physical and mental.
Mini-BEST Test (Balance Assessment Systems Test) | 15-20 minute
  Mini-BEST Test (Balance Assessment Systems Test) was used to evaluate the balance.
  Mini-BESTest is the shortest version of BESTest. Test include 4 subheading named preparatory movement, reactive postural control, sensory orientation and dynamic gait. Each subheading has its own total scoring. The total score of preparatory movement, reactive postural control and sensory orientation was 6, and the total score of the dynamic walking subheading was 10 points. The highest score in the test is 28.
  As the score decreases, the physical condition deteriorates. Each case tested has 3 points, 0-1-2, which are defined as severe, moderate and normal, respectively. One of these 3 points is selected based on the patient's performance in the tested condition.
The 5-repetition sit-to-stand test | 10 minute
  This test has been shown to provide information about lower extremity muscle strength in MS patients.
  The 5-repetition sit-to-stand test is a measure of the time taken to complete five repetitions of the sit-to-stand movement.

CONTACTS AND LOCATIONS:
Overall Officials: Nezire KÖSE, Prof., Principal Investigator — Hacettepe University; Rana KARABUDAK, Prof., Study Chair — Hacettepe University; Meryem A TUNCER, Prof., Study Chair — Haceetepe University; Kadriye ARMUTLU, Prof., Principal Investigator — Hacettepe University; Yeliz SALCI, Asts. Prof., Principal Investigator — Hacettepe University; Jale KARAKAYA, Assoc. Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Langeskov-Christensen M, Heine M, Kwakkel G, Dalgas U. Aerobic capacity in persons with multiple sclerosis: a systematic review and meta-analysis. Sports Med. 2015 Jun;45(6):905-23. doi: 10.1007/s40279-015-0307-x. PMID 25739555
- [Background] Skumlien S, Hagelund T, Bjortuft O, Ryg MS. A field test of functional status as performance of activities of daily living in COPD patients. Respir Med. 2006 Feb;100(2):316-23. doi: 10.1016/j.rmed.2005.04.022. Epub 2005 Jun 6. PMID 15941658
- [Background] Savci S, Inal-Ince D, Arikan H, Guclu-Gunduz A, Cetisli-Korkmaz N, Armutlu K, Karabudak R. Six-minute walk distance as a measure of functional exercise capacity in multiple sclerosis. Disabil Rehabil. 2005 Nov 30;27(22):1365-71. doi: 10.1080/09638280500164479. PMID 16372431
- [Background] Nicholl CR, Lincoln NB, Playford ED. The reliability and validity of the Nottingham Extended Activities of Daily Living Scale in patients with multiple sclerosis. Mult Scler. 2002 Oct;8(5):372-6. doi: 10.1191/1352458502ms827oa. PMID 12356202
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevoglu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Nottingham Extended Activities of Daily Living Scale. Aging Clin Exp Res. 2008 Oct;20(5):400-5. doi: 10.1007/BF03325144. PMID 19039280
- [Background] Moller AB, Bibby BM, Skjerbaek AG, Jensen E, Sorensen H, Stenager E, Dalgas U. Validity and variability of the 5-repetition sit-to-stand test in patients with multiple sclerosis. Disabil Rehabil. 2012;34(26):2251-8. doi: 10.3109/09638288.2012.683479. Epub 2012 May 22. PMID 22612360
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Idiman E, Uzunel F, Ozakbas S, Yozbatiran N, Oguz M, Callioglu B, Gokce N, Bahar Z. Cross-cultural adaptation and validation of multiple sclerosis quality of life questionnaire (MSQOL-54) in a Turkish multiple sclerosis sample. J Neurol Sci. 2006 Jan 15;240(1-2):77-80. doi: 10.1016/j.jns.2005.09.009. Epub 2005 Nov 8. PMID 16277993
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Cameron M, Mazumder R, Murchison C, King L. Mini Balance Evaluation Systems Test in people with multiple sclerosis: reflects imbalance but may not predict falls. Gait Posture. 2014;39(1):669. doi: 10.1016/j.gaitpost.2013.08.009. Epub 2013 Oct 17. No abstract available. PMID 24184138
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Mansson E, Lexell J. Performance of activities of daily living in multiple sclerosis. Disabil Rehabil. 2004 May 20;26(10):576-85. doi: 10.1080/09638280410001684587. PMID 15204511
- [Background] Marrie RA, Hanwell H. General health issues in multiple sclerosis: comorbidities, secondary conditions, and health behaviors. Continuum (Minneap Minn). 2013 Aug;19(4 Multiple Sclerosis):1046-57. doi: 10.1212/01.CON.0000433284.07844.6b. PMID 23917100
- [Background] Stickland MK, Butcher SJ, Marciniuk DD, Bhutani M. Assessing exercise limitation using cardiopulmonary exercise testing. Pulm Med. 2012;2012:824091. doi: 10.1155/2012/824091. Epub 2012 Nov 19. PMID 23213518
- [Background] Karloh M, Araujo CL, Gulart AA, Reis CM, Steidle LJ, Mayer AF. The Glittre-ADL test reflects functional performance measured by physical activities of daily living in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2016 Apr 8;20(3):223-30. doi: 10.1590/bjpt-rbf.2014.0155. PMID 27437713
- [Derived] Kaya G, Kose N, Salci Y, Armutlu K, Karakaya J, Tuncer A, Karabudak R. Reliability and validity of the glittre activities of daily living test in fully ambulatory multiple sclerosis patients. Ir J Med Sci. 2023 Oct;192(5):2379-2386. doi: 10.1007/s11845-022-03237-x. Epub 2022 Dec 1. PMID 36451004